CLINICAL TRIAL: NCT00406822
Title: Study of the Safety and Effectiveness of the OculusGen Collagen Matrix Implant as an Aid in Glaucoma Surgery
Brief Title: OculusGen-Glaucoma Historical Control Study in Taiwan
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to the change of supplier and sponsor
Sponsor: Pro Top & Mediking Company Limited (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mediking 0502
Record Dates: First submitted 2006-10-10; First posted 2006-12-04 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2007-06

CONDITIONS: Glaucoma
Keywords: Glaucoma; collagen matrix; OculusGen; trabeculectomy; tissue engineering
MeSH Terms: conditions — Glaucoma

INTERVENTIONS:
Device: OculusGen Biodegradable Collagen Matrix Implant

SUMMARY:
The purpose of this study is to determine whether the OculusGen Collagen Matrix are effective and safe to implant as an aid of glaucoma surgery.

DETAILED DESCRIPTION:
OculusGen® Collagen Matrix is a porous, scaffold matrix. It is to be implanted on the top of the scleral flap and beneath the conjunctiva and Tenon's capsule at the end of trabeculectomy. The pores in the scaffold matrix range from 20 to 200µm, a size that is suitable for fibroblasts to grow randomly, through the body of the matrix without causing scarring. The space occupied by the collagen matrix scaffold creates room for the development of a filtration bleb. Immediately after implantation, the collagen matrix is absorbed with the aqueous humor that bring a certain pressure press on the top of scleral flap which makes the dynamic balance for the aqueous system to keep the IOP in the right side. The collagen matrix is bio-degraded within 90 days and will leave a physiologic space for the filtration bleb to facilitate control of intraocular pressure (IOP).

ELIGIBILITY:
Subject inclusion criteria:

1. Age 18 years or over.
2. At least one eye diagnosed with glaucoma and receiving maximally tolerated medical therapy.
3. Subject able and willing to cooperate with investigation plan.
4. Subject able and willing to complete postoperative follow-up requirements.
5. Subject willing to sign informed consent form.

Subject exclusion criteria:

1. Have allergic reactions to collagen
2. Subject is taking anticoagulation and/or the physician does not suggested to stop taking the medication
3. Normal tension glaucoma patient
4. Subject has one eye received OculusGen™ implantation
5. Subject who been diagnosed infection with the operation eye
6. Subject with anterior chamber abnormality
7. Subject with steroid glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-12

PRIMARY OUTCOMES:
the effectiveness via the reduction of IOP | 180 day

SECONDARY OUTCOMES:
the safety via the incidence of complications and adverse events. | 180day

CONTACTS AND LOCATIONS:
Overall Officials: Henry SL Chen, MD, Principal Investigator — Chang Gung Memorial Hospital-Taipei Branch
Locations (1):
- Chang Gung Memorial Hospital -Taipei Branch, Taipei, Taiwan

REFERENCES:
- [Result] Hsu WC, Spilker MH, Yannas IV, Rubin PA. Inhibition of conjunctival scarring and contraction by a porous collagen-glycosaminoglycan implant. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2404-11. PMID 10937547